CLINICAL TRIAL: NCT04251858
Title: Evaluation of Oral Condition and the Effect of Dental Treatment on Physical Parameters of Athletes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Universidade Metropolitana de Santos (Other)
Responsible Party: Principal Investigator, CAIO VINICIUS G. ROMAN TORRES, Professor, Universidade Metropolitana de Santos
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SantosMU8
Record Dates: First submitted 2020-01-23; First posted 2020-02-05 (Actual); Last update posted 2021-05-24 (Actual); Status verified 2021-05

CONDITIONS: Periodontal Diseases; Inflammation Gum; Caries,Dental
Keywords: Periodontal Diseases; Athletes; Caries, dental; Periodontal index
MeSH Terms: conditions — Periodontal Diseases; Gingivitis; Dental Caries | interventions — Dental Scaling

STUDY DESIGN:
Intervention Model Description: The groups of participants should be divided by the oral condition of the participants (with oral problems and without oral problems)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Athletes with oral problems (Experimental): Athletes with periodontal diseases or gingivitis
  Interventions: Procedure: Dental Scaling; Other: Oral hygiene instruction
- Athletes without oral problems (No Intervention): Athletes diagnosed without oral problems

INTERVENTIONS:
Procedure: Dental Scaling — The individuals will be treated by a single periodontist and the scaling and root planing procedures will be performed on all teeth as follows: local anesthetic infiltrative type of the areas to be treated, dental and root scaling using Grace 5/6 carbon steel curettes, 11/12, 13/14 and MacCall 13/14, 17/18 curettes, according to their therapeutic indications. Polishing the quadrants treated with abrasive paste; oral hygiene instructions including Bass toothbrushing, dental floss and sometimes inter-dental brush.
  Arms: Athletes with oral problems
Other: Oral hygiene instruction — Oral hygiene instructions should be given to all study participants. Guidance on the most appropriate toothbrush, toothpaste and interproximal cleaning method.
  Arms: Athletes with oral problems

SUMMARY:
It is essential that athletes have perfect general health. Oral health plays an important role in this healthy framework necessary so that the results that must be achieved by athletes are not influenced. Inflammatory and / or infectious processes such as periodontal disease, caries, or even joint problems such as temporomandibular joint dysfunction can affect performance or impair participation in training and competitions.

DETAILED DESCRIPTION:
The objective of this longitudinal clinical study will be to evaluate the effect of dental treatment on individuals who practice physical activities through physical parameters of strength, speed and resistance. According to an initial survey, about 120 individuals should be examined. Clinical parameters such as decayed, lost and / or filled dental index and periodontal parameters such as probing depth (PS), clinical level of insertion (NCI), plaque index (IP) and bleeding index (IS) will be evaluated . Physical tests of strength, speed and resistance should be performed and periodontal therapy should be performed according to the needs presented by each individual. After 90 days, new clinical examinations and physical tests should be performed. The results obtained should be tabulated and analyzed. The investigators believe that individuals with oral inflammation / infection, the physical performance should be higher after performing periodontal therapy. Pro inflammatory cytokines present in high concentrations in the presence of periodontal disease can influence fatigue and difficulty in recovering from injuries, variables so important in an athlete's life.

ELIGIBILITY:
Inclusion Criteria:

* Athletes from all sports,
* Individuals with systemic pathologies, smokers, should be included in the study

Exclusion Criteria:

* pregnancy or lactation, use of antibiotics in the last 3 months, phenytoin, calcium antagonists, cyclosporine or anti-inflammatory drugs one month before the initial consultation, use of oral or replacement contraceptives hormonal, periodontal treatment in the 6 months prior to the start of the study.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-03-30 (Actual); Primary Completion 2020-11-10 (Actual); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Probing depth | 90 days
  Evaluation of Probing depth, from the gingival margin to the end of the periodontal sulcus
Clinical attachment level | 90 days
  evaluation of clinical attachment level, from the enamel cementum junction to the end of the periodontal sulcus
Gingival index | 90 days
  evaluation of bleeding on probing
Plaque index | 90 days
  evaluation of the accumulation of bacterial plaque around the teeth
DMF index | 90 days
  evaluation of teeth decayed, missed or filled
Aerobic running performance evaluation test | 90 days
  Run of 100 meters and time obtained in seconds and thousands of a second
critical speed in swimming | 90 days
  swim 25 meters, time measured in minutes and seconds
Body mass index | 90 days
  The BMI calculation must be done using the following mathematical formula: Weight ÷ height x height.
Muscle strength through the 1RM test on the bench press | 90 days
  It is the maximum amount of weight lifted once while performing a standardized weightlifting exercise. To test 1 RM of a muscle group, such as elbow flexors or knee extensors, a weight is chosen at the exercise device, but below the individual's maximum lifting capacity. If a repetition is completed, weight is added to the exercise device. Until the maximum lifting capacity is launched.
short-term heart rate variability at rest | 90 days
  To measure heart rate variability, we will use Polar S810i® frequency meter to obtain RR interval series for each individual, at rest, for 5 minutes; posteriorly, analysis will be performed using linear and non-linear indices.

CONTACTS AND LOCATIONS:
Overall Officials: CAIO VINICIUS G ROMAN TORRES, Principal Investigator — University of Santo Amaro
Locations (1):
- Caio Vinicius Gonçalves Roman Torres, Santos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] D'Ercole S, Tieri M, Martinelli D, Tripodi D. The effect of swimming on oral health status: competitive versus non-competitive athletes. J Appl Oral Sci. 2016 Apr;24(2):107-13. doi: 10.1590/1678-775720150324. PMID 27119757
- [Result] Needleman I, Ashley P, Meehan L, Petrie A, Weiler R, McNally S, Ayer C, Hanna R, Hunt I, Kell S, Ridgewell P, Taylor R. Poor oral health including active caries in 187 UK professional male football players: clinical dental examination performed by dentists. Br J Sports Med. 2016 Jan;50(1):41-4. doi: 10.1136/bjsports-2015-094953. Epub 2015 Nov 2. PMID 26527674
- [Result] Broad EM, Rye LA. Do current sports nutrition guidelines conflict with good oral health? Gen Dent. 2015 Nov-Dec;63(6):18-23. PMID 26545270

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-08-09): https://cdn.clinicaltrials.gov/large-docs/58/NCT04251858/Prot_SAP_000.pdf
  • Informed Consent Form (2018-08-09): https://cdn.clinicaltrials.gov/large-docs/58/NCT04251858/ICF_001.pdf